CLINICAL TRIAL: NCT03463707
Title: Multicenter, Double-blind, Randomized, Placebo-controlled Phase III Confirmatory Study of the Efficacy and Safety of BP101 in Female Patients With Decrease or Loss of Sexual Desire
Brief Title: BP101 for Adults With Female Sexual Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ivix LLX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP101-SD02-RUS
Record Dates: First submitted 2018-02-26; First posted 2018-03-13 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Hypoactive Sexual Desire Disorder; Female Sexual Dysfunction; Sexual Desire Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with BP101 (Experimental)
  Interventions: Drug: BP101
- Treatment with placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP101 — Investigational product BP101, nasal spray
  Arms: Treatment with BP101
Drug: Placebo — Placebo to Investigational product BP101, nasal spray
  Arms: Treatment with placebo

SUMMARY:
This study is to confirm efficacy and safety of study drug BP101 in female patients with with decrease or loss of sexual desire, which is equal to acquired generalized hypoactive sexual desire disorder (HSDD). Patients will be randomized in 1:1 ratio to either BP101 or placebo arms.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 21 to 50 years old, who have signed informed concent, with a regular menstrual cycle (STRAW stages -5 to -3).
* Decrease or loss of sexual desire (ICD-10 code: F-52.0) corresponding to the diagnosis of acquired generalized hypoactive sexual desire disorder (HSDD) according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM4), criteria.
* Current HSDD episode lasting not less than 24 weeks.
* Not less than 15 scores according to the FSDS-R (Distress) Total Score.
* Stable monogamous relationship with one sexually active male sexual partner lasting at least a year. The partner is physically available not less than 50% of time during a month.
* Consent to attempt to have a sexual intercourse at least twice a month, if she has a desire.
* Consent to complete a diary every day during the screening period and assessment of the baseline state (in this period diary records must cover ≥80% days), during the therapy and subsequent follow-up.
* Consent to use adequate methods of contraception throughout the study.

Exclusion Criteria:

* Any prohibited treatments.
* Other mental disorders or psychiatric diseases.
* Diagnosed Decrease or loss of sexual desire (HSDD) is situational (reactive) or lifelong.
* Score ≥ 20 according to the Beck Depression Inventory during the screening. Patients with 16 to 19 scores according to Beck's inventory may be included in the study unless, in the investigator's opinion, an actual depressive disorder is observed in the patient.
* Inflammatory diseases of pelvic organs, infections of the genitourinary system, cervicitis, interstitial cystitis, vulvodynia or severe atrophy of the vaginal epithelium, precluding normal sexual activity.
* Surgical interventions (other than cosmetic surgeries) on reproductive organs in past medical history (ovariectomy, hysterectomy, obvious scars from childbirth-related perineal stitches, etc), resulting in pain/dyspareunia, and/or precluding sexual contacts, and/or requires hormonal replacement treatment, and/or lead to the loss of sensibility while sexual contact.
* Pregnant and nursing women or non-lactating women during the first 12 months after childbirth.
* Consumption of more than 5 portions of alcoholic drinks per week or alcohol addiction, drug addiction or drug abuse in the past. One portion of an alcoholic drink means 360 ml of beer, 120 ml of wine or 30 ml of a strong alcoholic drink.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged from 21 to 50 years old
Enrollment: 205 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Satisfying sexual events | Baseline and 4 weeks of treatment
  Change in the number of satisfying sexual events (SSEs), standardized to the 28-day period, after 4 weeks of treatment, compared with the baseline.

SECONDARY OUTCOMES:
Satisfying sexual events | Baseline and 4 and 8 weeks of follow-up
  Change in the number of satisfying sexual events (SSEs), standardized to the 28-day period, after 4 and 8 weeks of follow-up, compared with the baseline.
Orgasms | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the number of orgasms, standardized to the 28-day period, after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
Female Sexual Function Index total score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function Index (FSFI) total score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSFI total score ranges from 2.0 to 36.0, where higher score represents better sexual function. FSFI total score is a sum of FSFI individual domains scores (individual domains are: Desire, Arousal, Lubrication, Orgasm, Satisfaction, and Pain).
Female Sexual Function Index Desire domain score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function Index (FSFI) Desire domain score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSFI Desire domain score ranges from 1.2 to 6.0, where higher score represents better sexual desire.
Female Sexual Function Index Arousal domain score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function Index (FSFI) Arousal domain score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSFI Arousal domain score ranges from 0 to 6.0, where higher score represents better sexual arousal.
Female Sexual Function Index Lubrication domain score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function Index (FSFI) Lubrication domain score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSFI Lubrication domain score ranges from 0 to 6.0, where higher score represents better vaginal lubrication.
Female Sexual Function Index Orgasm domain score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function Index (FSFI) Orgasm domain score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSFI Orgasm domain score ranges from 0 to 6.0, where higher score represents better orgasm sensation.
Female Sexual Function Index Satisfaction domain score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function Index (FSFI) Satisfaction domain score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSFI Satisfaction domain score ranges from 0.8 to 6.0, where higher score represents better sexual satisfaction.
Female Sexual Function Index Pain domain score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function Index (FSFI) Pain domain score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSFI Pain domain score ranges from 0 to 6.0, where higher score represents lower pain sensation during sexual intercourse.
Female Sexual Distress Scale-Revised Total score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Distress Scale-Revised (FSDS-R) total score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSDS-R total score ranges from 0 to 52, where higher score represents higher level of distress related to sexual activities. A score of ≥11 discriminates between women with female sexual disfunction (score of ≥11) and no female sexual disfunction (score of <11).
Female Sexual Distress Scale-Revised Item 13 score | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Distress Scale-Revised (FSDS-R) Item 13 score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSDS-R Item 13 score ranges from 0 to 4, where higher score represents higher level of bother by low sexual desire.
Sexual function according to the Female Sexual Function questionnaire | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  Change in the Female Sexual Function questionnaire (FSF) score after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
  FSF score ranges from 0 to 36, where higher score represents better sexual function.
Patient's assessment of efficacy of the therapy according to the Patient Global Impression of Improvement | Baseline and 4 weeks of treatment, 4 and 8 weeks of follow-up
  The patient's assessment of efficacy of the therapy according to the Patient Global Impression of Improvement (PGI-I) after 4 weeks of therapy and after 4 and 8 weeks of follow-up, compared with the baseline.
Number of adverse events | During 12 weeks after start of treatment (4 weeks of treatment and 8 weeks of follow-up)
  Frequency of adverse events reporting, including serious adverse events, in treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniil G. Nemenov, MD, Study Director — Ivix LLX
Locations (20):
- Russia (20):
  - Алтайский государственный медицинский университет, Barnaul
  - Kazan State Medical University, Kazan'
  - Kuban State Medical University, Krasnodar
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - N.A. Alexeev Moscow Psychiatric Clinical Hospital #1, Moscow
  - National Medical Research Center of Obstetrics, Gynecology and Perinatology, Moscow
  - National Medical Research Center of Psychiatry and Addiction named after V.P. Serbsky, Moscow
  - Clinical Psychiatry Hospital №1, Nizhny Novgorod
  - Orenburg Regional Clinical Psychiatric Hospital No. 2, Orenburg
  - City psychiatric hospital №7 named after academician I.P. Pavlov, Saint Petersburg
  - Doctor SAN Ltd., Saint Petersburg
  - Leningrad Regional Narcological Dispensary, Saint Petersburg
  - OrKli Hospital LLC, Saint Petersburg
  - Research center Eco-Safety LLC, Saint Petersburg
  - Samara Psychiatric Hospital, Samara
  - Regional Clinical Psychiatric Hospital of St. Sofia, Saratov
  - Engels Psycyatric hospital, Saratovskaya
  - Clinic "Hundred Years", Tomsk
  - Bashkir State Medical University, Ufa
  - Yaroslavl Regional Clinical Psychiatric Hospital, Yaroslavl

IPD SHARING:
Plan to Share IPD: No